CLINICAL TRIAL: NCT02165059
Title: Indiana University GI Neuromuscular Pathology Prospective Registry
Brief Title: GI Neuromuscular Pathology Prospective Registry
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John M. Wo, MD, Indiana University
Other Study IDs: GI Neuromuscular Pathology
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Gastroparesis
Keywords: Nausea; Vomiting; Functional dyspepsia; Bloating; Regurgitation; Retching
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting; Gastroesophageal Reflux | interventions — Biopsy; Surgical Procedures, Operative; Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Full thickness biopsies of Gastric body and proximal jejunum obtained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GI Neuromuscal Disorder Cohort: Patients who are undergoing surgical full-thickness biopsy of the stomach and/or proximal jejunum for the clinical evaluation of GI neuromuscular disorder
  Interventions: Procedure: Surgical Full Thickness Biopsy
- GI Surgery Patients without neuromuscal disorders (control) cohort: Patients undergoing esophagectomy, sleeve gastrectomy for obesity, Roux-en-Y gastric bypass, whipple surgery, transplant surgery, or organ donors.
  Interventions: Procedure: Surgical Full Thickness Biopsy

INTERVENTIONS:
Procedure: Surgical Full Thickness Biopsy — Eligible subjects will undergo a surgical full thickness biopsy of the stomach and/or proximal jejunum as part of their planned surgery.
  Other Names: Biopsy; Surgical; Full-thickness; Stomach

SUMMARY:
In this research study, biopsy samples will be collected to provide more insight into the underlying cause of the motility disorders, help direct further investigation into the cause of the underlying condition, provide future prognosis and predict response to gastric electrical stimulation (GES).

DETAILED DESCRIPTION:
Biopsies will be collected from patients that have been diagnosed with gastroparesis (having nausea, retching, bloating and fullness of stomach) and are undergoing surgery for the GES implantation. These patients will serve as our study group population. Biopsy samples of those who do not have gastroparesis but are undergoing surgery on the digestive system will be collected after the patients consent to be on the trial. These patients will serve as our control group population. Detailed medical history will be collected and the study group patients will be asked to complete two questionnaire to assess the severity of the symptoms. They will be followed in the clinic at 6, 12, 18 and 24 months post implantation.

ELIGIBILITY:
Inclusion Criteria Study Group:

Patients who are undergoing surgical full-thickness biopsy of the stomach and/or proximal jejunum for the clinical evaluation of GI neuromuscular disorder.

Inclusion Criteria Control Group:

Patients undergoing esophagectomy, sleeve gastrectomy for obesity, or Roux-en Y gastric bypass Patients undergoing Whipple surgery Patients undergoing transplant surgery

Patients who are organ donors and undergoing surgery

Exclusion Criteria Study Group:

Contraindication for surgical full-thickness biopsy for any reason. Significant comorbidity due to severe cardiovascular, renal, pulmonary, or liver disease.

Significant coagulopathy Non-ambulatory patients: bed-ridden, nursing home resident. Pregnant Unable to give own informed consent Prisoners

Exclusion Criteria Control Group:

Prior diagnosis of gastroparesis Prior diagnosis of chronic intestinal pseudo-obstruction Unable to give own informed consent if not an organ donor

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with gastropareiss and are undergoing surgery for full thickness biopsy GES implantation willl serve as our study group, Patients who are undergoing surgery on the digestive system but do not have gastroparesis, will serve as our control group.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biologic Markers As Predictors for Gastric Electrical Stimulation Outcomes | from implantation to 6 months after
  To determine if ICC abnormalities of the stomach and proximal jejunum can be used as a biologic marker in predicting clinical outcome in patients undergoing surgical implantation of gastric electrical stimulation (GES) for severe gastroparesis.

CONTACTS AND LOCATIONS:
Overall Officials: John M Wo, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hosptial, Indianapolis, Indiana, United States